CLINICAL TRIAL: NCT00311857
Title: Treatment of Primary Glioblastoma Multiforme With Cetuximab, Radiotherapy and Temozolomide (GERT) - Phase I/II Trial
Brief Title: Safety Study of Cetuximab, Radiotherapy and Temozolomide in Primary Glioblastoma Multiforme(GERT)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudract-2005-003911-63; PEI 119/01
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Glioblastoma Multiforme
Keywords: Cetuximab
MeSH Terms: conditions — Glioblastoma | interventions — Cetuximab; Temozolomide; Radiotherapy

INTERVENTIONS:
Drug: Cetuximab
Drug: Temozolomide
Procedure: Radiation therapy

SUMMARY:
GERT is a one-armed single-center phase I/II trial. In a first step, dose-escalation of TMZ from 50 mg/m2 to 75mg/m2 together with radiotherapy and cetuximab will be performed. Should safety be proven, the phase II trial will be initiated with the standard dose of 75mg/m2 of TMZ. Cetuximab will be applied in the standard application dose of 400mg/m2 in week 1, thereafter at a dose of 250mg/m2 weekly. A total of 46 patients will be included into this phase I/II trial.

Primary endpoints are feasibility and toxicity, secondary endpoints are overall and progression-free survival. An interim analysis will be performed after inclusion of 15 patients into the main study. Patients' enrolment will be performed over a period of 2 years. The observation time will end 2 years after inclusion of the last patient.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 and < 70 years of age
* Karnofsky Performance Score >= 60
* histologically confirmed supratentorial GBM
* interval between primary diagnosis and registration for the study < 4 weeks
* patients will be included according to the incidental gender distribution for patients with GBM of ♀/♂ 2:3
* adequate blood values (not older than 14 days prior to initiation of RCHT)
* neutrophil count (ANC) ≥1500/mm3 or white blood cells (WBC) ≥2000/mm3
* platelets ≥100.000/mm3
* hemoglobin ≥10g/dL
* BUN <1.5 times the upper range
* Total and direct bilirubin <1.5times the upper laboratory limit
* Adequate liver enzymes <3 times the upper laboratory limit
* Life expectancy >12 weeks
* Written informed consent

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy of the brain or chemotherapy with DTIC or TMZ
* known allergy against extrinsical proteins
* previous chemotherapy or therapy with an EGFR-inhibitor
* Previous antibody therapy
* Patients who have not yet recovered from acute toxicities of prior therapies
* Acute infections requiring systemic application of antibiotics
* Frequent vomiting or a medical condition preventing the oral application of TMZ
* Clinically active kidney- liver or cardiac disease
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin)
* HIV
* Pregnant or lactating women
* Participation in another clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2006-02

PRIMARY OUTCOMES:
Toxicity

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Schulz-Ertner, MD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany